CLINICAL TRIAL: NCT00986544
Title: Drain After Elective Laparoscopic Cholecystectomy. A Randomized Controlled Trial
Brief Title: Drain After Elective Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Erasmo Spaziani, MD; PhD, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pic63
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Results first posted 2012-03-23 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-02

CONDITIONS: Cholelithiasis
Keywords: Laparoscopy; cholecystectomy; drainage
MeSH Terms: conditions — Cholelithiasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Absence of drain (Sham Comparator)
  Interventions: Procedure: no drain; Procedure: drain not positioned
- Drain (Active Comparator): drain positioned in the subhepatic space after laparoscopic cholecystectomy
  Interventions: Procedure: drain positioned

INTERVENTIONS:
Procedure: no drain — drain positioned on the skin
  Arms: Absence of drain
Procedure: drain positioned — drain positioned in the subhepatic space
  Arms: Drain
Procedure: drain not positioned — Drain positioned in the abdominal wall
  Arms: Absence of drain

SUMMARY:
The trial aims to assess the value of drains in elective laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
After laparoscopic gallbladder removal patients are randomized to have a suction drain positioned in the subhepatic space or to have a sham drain in the subhepatic space. The primary outcome measure will be the presence of subhepatic fluid collection at ultrasonographic examination on the first postoperative day. Secondary outcome measures will be postoperative abdominal and shoulder tip pain, use of analgesics, nausea, vomiting and morbidity

ELIGIBILITY:
Inclusion Criteria:

* elective laparoscopic cholecystectomy

Exclusion Criteria:

* acute cholecystitis, cholangitis, or pancreatitis
* no contraindication for the laparoscopic
* no other additional procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2009-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erasmo Spaziani, PhD, Study Director — University of Rome "La Sapienza"- Polo Pontino
Locations (1):
- University of Rome "La Sapienza" - Polo Pontino, Terracina, Latina, Italy

REFERENCES:
- [Background] Gurusamy KS, Samraj K, Mullerat P, Davidson BR. Routine abdominal drainage for uncomplicated laparoscopic cholecystectomy. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD006004. doi: 10.1002/14651858.CD006004.pub3. PMID 17943873
- [Background] Tzovaras G, Liakou P, Fafoulakis F, Baloyiannis I, Zacharoulis D, Hatzitheofilou C. Is there a role for drain use in elective laparoscopic cholecystectomy? A controlled randomized trial. Am J Surg. 2009 Jun;197(6):759-63. doi: 10.1016/j.amjsurg.2008.05.011. Epub 2008 Oct 16. PMID 18926516

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From December 1, 2009 to December 31, 2010 patients were submitted to laparoscopic cholecystectomy in Hospital "P.Colombo", Velletri, Italy; University of Rome "La Sapienza"- Polo Pontino, Terracina, Italy; Obafemi Awolowo University, Ile-Ife, Nigeria.
Pre-assignment Details: Patients with acute cholecystitis, cholangitis, or pancreatitis were excluded. If intraoperative common bile duct exploration or any other additional procedure were performed, patients were also excluded
Groups:
- Absence of Drain: After laparoscopic gallbladder removal no suction drain positioned in the subhepatic space.
Period: Overall Study
Arm/Group | Absence of Drain | Drain
Started | 53 | 53
Completed | 53 | 53
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Absence of Drain | Drain | Total
Number analyzed (Participants) | 53 | 53 | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 34 | 72
  >=65 years | 15 | 19 | 34
Age Continuous [Mean (Standard Deviation); unit: years] | 47.1 (16.7) | 48.6 (14.2) | 47.8 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 42 | 82
  Male | 13 | 11 | 24
Region of Enrollment [Number; unit: participants]
  Italy | 53 | 53 | 106

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Subhepatic Collection at Ultrasonographic Examination
Description: An abdominal ultrasonography was routinely performed on the first postoperative day with the aim to detect any fluid collection. If present, the volume in ml of subhepatic collection was calculated.
Time Frame: first postoperative day
Population: An intention to treat (ITT) analysis was performed.
Measure: Number; unit: Participants
Arm/Group | Absence of Drain | Drain
Number analyzed (Participants) | 53 | 53
Participants | 45 | 46

2. Secondary Outcome: Number of Participants With Postoperative Complications
Time Frame: 1 month
Population: Intention to treat analysis
Measure: Number; unit: participants
Arm/Group | Absence of Drain | Drain
Number analyzed (Participants) | 53 | 53
participants | 3 | 4

ADVERSE EVENTS:
Arm/Group | Absence of Drain | Drain
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/53
Other Adverse Events (participants affected / at risk) | 0/53 | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No